CLINICAL TRIAL: NCT02449148
Title: Healthy Nutrition and Energy Restriction as Cancer Prevention Strategies: a Randomized Controlled Intervention Trial
Brief Title: Nutrition and Energy Restriction for Cancer Prevention
Acronym: HELENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Tilman Kuehn, Dr. Tilman Kühn, German Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DKFZ Study_ID 670
Record Dates: First submitted 2015-04-01; First posted 2015-05-20 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Visceral Obesity; Weight Loss; Metabolic Diseases; Body Composition, Beneficial
Keywords: energy restriction; fasting; intermittent fast; cancer prevention; subcutaneous fat tissue gene expression
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Weight Loss; Metabolic Diseases; Glucocorticoid Receptor Deficiency; Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intermittent Calorie Restriction (Experimental): 2 days per week fasting with 25 % energy intake and 5 days per week at 100% energy intake
  Interventions: Other: Calorie Restriction
- Continuous Calorie Restriction (Experimental): daily energy intake of 80 %
  Interventions: Other: Calorie Restriction
- Healthy Nutrition (No Intervention): general advice on healthy nutrition

INTERVENTIONS:
Other: Calorie Restriction — diet intervention to reduce the risk for obesity associated diseases
  Other Names: weight loss trial;
  Arms: Continuous Calorie Restriction; Intermittent Calorie Restriction

SUMMARY:
This study evaluates the effect of intermittent calorie restriction versus continued calorie restriction on weight loss, gene expression profile of subcutaneous adipose tissue and abdominal fat distribution.

DETAILED DESCRIPTION:
Since obesity has become a major public health concern appropriate strategies are needed in order to reduce obesity-related health risks in later life span. Obesity is one of the main risk factors not only for diabetes and cardiovascular diseases, but also for several types of cancer. Several key mechanisms, which may link obesity, metabolic dysregulation and cancer risk, such as obesity-driven inflammation, altered adipokine, growth factor and sex hormone signaling, and changes in the microbiota have been identified.

Various studies have shown that continuous calorie restriction (CCR) and exercise are effective strategies to enforce weight-loss and improve biomarker profiles. Intermittent calorie restriction (ICR) as a novel strategy might induce favorable metabolic changes and lead to higher compliance rates. The concept of this diet regime is very simple e.g. 2 days/week of fasting following a standardized diet covering 25 % of energy needs and 5 days/week of ad libitum consumption. To verify the effectiveness of ICR as an alternative weight loss strategy to CCR controlled intervention trials are required. Although both CCR and ICR induce a negative energy balance, the metabolic effect on human physiology might differ.

Within the HELENA-study 50 non-smoking adults (men and women aged 35 to 65 years) with an BMI ≥ 25 kg/m² and ≤ 40 kg/m² will be randomly assigned to each of the intervention arms: (1) ICR arm (2 day/week fasting, i.e. 25% energy intake, energy intake of 100% on 5 days/week leading to a weekly average energy intake of ~80%) (2) CCR arm (daily energy intake of 80%) and 3) control arm (general advice on healthy nutrition).

The trial will last 1 year, with an intervention phase of 12 weeks (weeks 0-12; intervention; close contact with participants), followed by a maintenance phase (weeks 13-24; maintenance; regular, but less frequent contact with participants) and a follow-up phase (weeks 25-52).

Biological specimens will be collected as follows:

Baseline (T0, week 1): Blood, urine, stool and subcutaneous adipose tissue samples; After 3 months (T1, week 13): Blood, urine, stool and subcutaneous adipose tissue samples; After 6 months (T2, week 25): Blood, urine, and stool; After 12 months (T3, week 52): Blood and urine; Magnet resonance tomography imaging (MRI, at T0, T1 and T3) and lifestyle assessments (nutrition behavior, physical activity and quality of life, T0-T3) will be performed to unravel the link to fat distribution, metabolic changes, health and lifestyle. The primary objective of the three-arm randomized controlled intervention trial is to investigate the effect of nutrition intervention on body weight and gene expression profile in subcutaneous adipose tissue of overweight and obese individuals. We hypothesize that better compliance rates will be achieved by the ICR rather than by the CCR group and that ICR will show a higher sustainability with respect to weight loss, weight maintenance, and biomarker profiles. The purpose of this study is further to analyze if the nutrition interventions and associated weight loss have different effects on abdominal fat distribution and liver fat content.

The statistical analysis will be carried out by using the SAS statistical software [SAS Institute Inc., Cary, NC, USA] or comparable software. Descriptive statistics, correlations and univariate analyses will be used to get insight on general characteristics of participants in the intervention groups. For the primary objective, two sided t-test and ANCOVA modelling will be performed to investigate whether changes in gene expression levels are affected by nutrition intervention. Comparisons between two groups (e.g. ICR and CCR or CCR/ICR and control group) will be carried out using t-tests and parallel comparison across the three groups will be carried out using ANCOVA models. Where applicable, the analyses will include adjustments for confounders, specially age and gender. Likewise, stratified analysis will be carried out as necessary. ANCOVA models will be performed to evaluate the effects of nutrition intervention on biomarker profiles, adjusted by strata age and gender. Similar evaluations will be performed for fat distribution patterns, quality of life, physical activity and nutrition patterns. In addition, correlation and linear regression analyses will be performed to measure effects of weight-loss, gene expression levels and metabolic profiles, controlled by nutrition intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 35 to 65 years
* Overweight or obese (BMI ≥ 25 kg/m2 ≤ 40 kg/m2 )
* German speaking
* Non- smoker
* Provision of written informed consent

Exclusion Criteria:

* Not able to understand and sign the informed consent form in person
* Already diagnosed diabetes
* HbA1c ≥ 6.5 % and/or fasting plasma glucose > 125 mg/dl
* History of cancer within the past 10 years
* Risk of bleeding disorders (e.g. Marcumar intake)
* Current or history of eating disorders (bulimia, anorexia, binge-eating)
* Pregnant or lactating during the past 12 months
* Increased or decreased thyroid-stimulating hormone in baseline blood check
* Already diagnosed hepatic dysfunction and/or increased or decreased γ-GT, GPT and/or GOT in baseline blood check
* Already diagnosed kidney dysfunction and/or increased or decreased creatinine, urea and/or uric acid in baseline blood check
* Medications that might affect the endpoints of the study e.g. immunosuppressive medication (cortisol, antibody treatment), hormone replacement therapy, medication for fat metabolism (e.g. statine, fibrate)
* Participation in another intervention study shorter than three months ago

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in subcutaneous adipose tissue measured by whole genome sequencing | Assessments at baseline (week 0), and after the intervention phase (week 13)

SECONDARY OUTCOMES:
Changes in abdominal fat distribution pattern (visceral, subcutaneous, total adipose tissue) measured by magnetic resonance spectroscopy | Assessments at baseline (week 0), after the intervention phase (week 13),and after the follow-up phase (week 52)
Changes in blood-based biomarkers, i.e. parameters of inflammation, adipokines, growth and hormonal factors, which have been shown to be associated with obesity-related chronic diseases before | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintenance phase (week 25), and after the maintenance phase (week 25)
Changes in weight (kg) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in BMI (kg/m2) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in waist circumference (cm) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in hip circumference (cm) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in blood pressure (mm/Hg) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in pulse (bpm) | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
Changes in quality of life (as defined by changes in SF-12-derived scores) | Assessments at baseline (week 0) and after the intervention phase (week 13)
Changes in liver fat content measured by magnetic resonance spectroscopy | Assessments at baseline (week 0), after the intervention phase (week 13),and after the follow-up phase (week 52)

OTHER OUTCOMES:
Changes in the composition of the gut microbiota by taxonomic, functional, and comparative analysis of sequencing data | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
  Exploratory Outcome
Changes in blood metabolites, as measured by LC-MS/MS-based targeted and untargeted metabolomics tools | Assessments at baseline (week 0), after the intervention phase (week 13), after the maintencance phase (week 25) and after the follow-up phase (week 52)
  Exploratory Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Kühn, PhD, Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Sowah SA, Milanese A, Schubel R, Wirbel J, Kartal E, Johnson TS, Hirche F, Grafetstatter M, Nonnenmacher T, Kirsten R, Lopez-Nogueroles M, Lahoz A, Schwarz KV, Okun JG, Ulrich CM, Nattenmuller J, von Eckardstein A, Muller D, Stangl GI, Kaaks R, Kuhn T, Zeller G. Calorie restriction improves metabolic state independently of gut microbiome composition: a randomized dietary intervention trial. Genome Med. 2022 Mar 14;14(1):30. doi: 10.1186/s13073-022-01030-0. PMID 35287713
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Schubel R, Nattenmuller J, Sookthai D, Nonnenmacher T, Graf ME, Riedl L, Schlett CL, von Stackelberg O, Johnson T, Nabers D, Kirsten R, Kratz M, Kauczor HU, Ulrich CM, Kaaks R, Kuhn T. Effects of intermittent and continuous calorie restriction on body weight and metabolism over 50 wk: a randomized controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):933-945. doi: 10.1093/ajcn/nqy196. PMID 30475957